CLINICAL TRIAL: NCT04120064
Title: Treatment of Vitamin D Deficiency With Large Bolus Cholecalciferol in the Outpatient Setting
Brief Title: Treatment of Vitamin D Deficiency With Large Bolus Cholecalciferol
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Covid19, not able to finish recruitment
Sponsor: Parkview Medical Center (Other)
Responsible Party: Principal Investigator, Doug Duffee, Administrator, Parkview Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIRB64
Record Dates: First submitted 2019-09-06; First posted 2019-10-09 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Large bolus (Experimental)
  Interventions: Drug: Cholecalciferol
- Standard (Active Comparator)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Large, one time dose of 300,000 IU oral cholecalciferol or daily 5,000 IU oral cholecalciferol

SUMMARY:
Comparing two treatment regimens (solitary large dose vs daily smaller dose) in patients diagnosed with vitamin D deficiency.

DETAILED DESCRIPTION:
Study is looking at patients with diagnosed vitamin D deficiency (<20ng/mL). Participants are healthy adults between 18 and 75. No diagnosis of cancer, pregnancy, hypercalcemia, hyperparathyroidism, gastrointestinal absorption disorder, or chronic kidney disease and not taking medications for seizures or osteoporosis. Participants are randomized into two treatment groups: (1) 5,000IU cholecalciferol daily or (2) one-time 300,000 international units (IU) cholecalciferol. Vitamin D level, calcium level, and renal function are measure one week after initiating treatment and then at 3 months, 6 months, 9 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75yrs old
* serum 25(OH)-vitamin D level <20ng/mL
* patient of Parkview Adult Medicine clinic
* not currently on cholecalciferol >2,000IU daily
* no ergocalciferol administration within last week

Exclusion Criteria:

* history of hypercalcemia or hyperparathyroidism
* history of chronic kidney disease with baseline creatinine >1.1
* history of gastric absorption abnormalities
* history of Paget's disease or osteomalacia
* history of thyrotoxicosis
* known malignancy
* currently pregnant
* taking medications for osteoporosis or seizures
* taking more than 1200mg/day of calcium
* inpatient hospitalization at the initiation of study meds

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment of vitamin D deficiency over a one year time frame: normalization of vitamin D levels above 30ng/mL | 12months
  Looking for normalization of vitamin D levels

SECONDARY OUTCOMES:
Duration of efficacy after starting vitamin D replacement as monitored at one week and then three month intervals for one year | 1 week, 3 months, 6 months, 9 months, 12 months
  Evaluation of how long participants maintain normal vitamin D levels with treatment
Compliance with therapy as measured by the reported number of missed doses at one week on therapy and then every three months for a year | 1 week, 3 months, 6 months, 9 months, 12 months
  Evaluation of missed doses

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Murphy, DO, Study Chair — Parkview Medical Center
Locations (1):
- Parkview Medical Center, Pueblo, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT04120064/Prot_000.pdf
  • Informed Consent Form (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT04120064/ICF_001.pdf